CLINICAL TRIAL: NCT02711982
Title: Clinical Treatment of Traumatic Optic Neuropathy: Optic Nerve Decompression Randomized Controlled Study
Brief Title: Surgery for Traumatic Optic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Hou Lijun, Professor, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016TON Study
Record Dates: First submitted 2016-03-06; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Optic Neuropathy
MeSH Terms: conditions — Optic Nerve Injuries | interventions — Methylprednisolone; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optic nerve decompression (Active Comparator): Optic canal and optic nerve sheath decompression within 5 days from trauma occur.
  Interventions: Procedure: Optic canal and optic nerve sheath decompression
- methylprednisolone (Active Comparator): a maximum daily dose of 1 g of methylprednisolone
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Procedure: Optic canal and optic nerve sheath decompression — within 5 days from trauma
  Other Names: optic decompression
  Arms: Optic nerve decompression
Drug: methylprednisolone — within 5 days from trauma
  Other Names: steroids
  Arms: methylprednisolone

SUMMARY:
The pathophysiology of Traumatic Optic Neuropathy (TON) include a primary and secondary mechanism of injury. At present, no studies validate a particular approach to the management of TON. There are three management lines for these patients that include 1)observation only;2)medical treatment with high or megadoses of methylprednisolone; and 3)surgical intervention. Studies have shown that forces applied to the frontal bone and malar eminences are transferred and concentrated in the area near the optic canal. The tight adherence of the optic nerve's dural sheath to the periosteum within the optic canal is also thought to contribute to this segment of the nerve being extremely susceptible to the deformative stresses of the skull bones. In this study, investigators aim to make a randomized controlled trial to certify the efficiency of optic nerve canal decompression for TON patients.

DETAILED DESCRIPTION:
surgical intervention's efficiency and outcome for TON patients will be clearly present after this randomized controlled trial study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the history of Traumatic Brain Injury or Craniofacial Trauma
* Optic nerve compression（intraneural edema, nerve sheath hematoma or canal fracture with impingement)
* Amplitude and latency abnormal or Ratio of amplitude of abnormal to normal side.

Exclusion Criteria:

* Glasgow Coma Scale，Score<8
* Patients with good Visual Acuity and Visual Evoked Potential amplitude ratio more than 50%
* Other Contraindications for surgery

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2010-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Amplitude and Latency of Visual-Evoked Potential | from trauma day to 60 days after trauma
  Name of Scale: Visual-Evoked Potential Physiological Parameter: Amplitude and Latency Questionnaire: Trauma day and 1 day, 2 days, 3 days, 7 days, 14 days, 30 days and 60 days after trauma. Two more test for the day before surgery（Medical） and the day after surgery(Medical).
  Measurement collection: Inpatient and outpatient

SECONDARY OUTCOMES:
Vision level of Visual Acuity | from trauma day to 60 days after trauma
  Name of Scale: Level Vision and Visual acuity chart from 0.1 to 1.5 Physiological Parameter: light perception, hand motion and Visual Acuity Chart from 0.1 to 1.5 Questionnaire: Trauma day and 1 day, 2 days, 3 days, 7 days, 14 days, 30 days and 60 days after trauma. Two more test for the day before surgery（Medical） and the day after surgery(Medical).
  Measurement collection: Inpatient and outpatient

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Hou, MD,PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Department of Neurosurgery,ShangHai ChangZheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No